CLINICAL TRIAL: NCT06614400
Title: MonitoRing the Effect of TRAnscutaneous Functional electrIcal Stimulation of the Common Peroneal Nerve on Cerebral Haemodynamics in Patients With Ischaemic Strokes. A Single Centre Prospective Study (Phase 1).
Brief Title: The RETRAIN Trial (Phase 1)
Acronym: RETRAIN
Status: Completed | Type: Observational
Sponsor: Countess of Chester NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 343056
Record Dates: First submitted 2024-08-28; First posted 2024-09-26 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Ischaemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objective is to investigate in stroke patients the impact of geko™ NMES treatment, when used as standard of care for VTE prevention, on brain haemodynamics at different stimulation levels and in three different postural positions (supine, semi-supine [45° seated] and seated). The aim is to identify the optimal stimulation level and postural position for the maximum response (NMES versus no NMES) with regard to relative total haemoglobin concentration (i.e., the sum of relative deoxyhaemoglobin and oxyhaemoglobin concentrations) using fNIRS and EEG.

ELIGIBILITY:
Inclusion Criteria:

* Adult over 18
* Patient with ischaemic stroke diagnosis confirmed by a stroke physician.
* No intracerebral haemorrhage as ruled out by computerised tomography (CT) or MRI scan.
* Able to achieve a supine, sitting and semi-sitting position of 45° with the help of another person.
* Receiving geko™ NMES treatment as standard of care for VTE prevention

Exclusion Criteria:

* Inability to gain consent from the patient.
* A transient ischaemic attack (TIA).
* Stroke survivors with ischaemic stroke less than 7 days from onset.
* History of epilepsy.
* Below/above knee amputation.
* History of established peripheral neuropathy.
* Too unwell to participate as judged by physician.
* Use of any other neuromodulation device that may interact with NMES

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (over 18 years) with ischaemic stroke more than 7 days from onset
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2024-10-08 (Actual); Primary Completion 2025-03-08 (Actual); Study Completion 2025-03-18 (Actual)

PRIMARY OUTCOMES:
Primary outcome | 3 hours
  a change in brain haemodynamics (or blood flow) in terms of oxygenated and de-oxygentated blood from baseline to end of study participation.

SECONDARY OUTCOMES:
Secondary objective | 3 hours
  Neurovascular coupling, Cerebral autoregulation and dynamic functional connectivity

CONTACTS AND LOCATIONS:
Locations (1):
- Countess of Chester Hospital NHS Foundation Trust, Chester, Cheshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
No identifiable patient data will be shared, only the findings of the procedure.